CLINICAL TRIAL: NCT04108767
Title: Innovative and Transdisciplinary Observation Program for the Quality of Life of Health Students
Acronym: POSITIVE
Status: Withdrawn | Type: Observational
Why Stopped: We were not able to conduct this study, in fact we opened the participating center and the confinement arrived a few days later. Since then, the organization of the students' follow-up has changed and made the study as it was thought obsolete.
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL19_0398
Record Dates: First submitted 2019-09-26; First posted 2019-09-30 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Healthy
MeSH Terms: interventions — Quality of Life; Health

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Health students enrolled in the 3rd year at the University Cla: Health students enrolled in the 3rd year at the University Claude Bernard Lyon 1, aged over 18 years.
  Interventions: Behavioral: Answer to standardized questionnaires in quality of life, health, lifestyle and behaviors

INTERVENTIONS:
Behavioral: Answer to standardized questionnaires in quality of life, health, lifestyle and behaviors — The cross-sectional study will be conducted in all students in health sciences in 3rd year enrolled at the University Claude Bernard Lyon 1 (UCBL) and participating at the required medical consultation at the college Health Department of UCBL, over a period of 9 months.
  The self-questionnaires will be completed by the students during the mandatory medical preventive visit at the university health center.
  All dimensions investigated by the questionnaire are usually questioned by the caregivers during the consultation as part of the usual follow-up of students.

SUMMARY:
Scientific context: Students' quality of life reflects the general health of students, in connection with the studies themselves, but also with physical, biological, social, cultural, and psychological determinants. Indeed, students are young adults exposed to a complex period composed of transitions in different spheres of their life: housing, domestic tasks, social learning, lifestyle choices, etc. In addition to this, students in medical and health sciences have to face with stress due to a demanding training and exposure to the hospital world. According to the Haute Autorité de Santé (HAS), health professionals in activity or in training are identified as a "population at risk historically identified."

The studies on stress and psychological disorders, in medical students, are considerably documented on the international level and the incidence of various psychic problems (depressive state, suicidal ideas ...) and behavioural (food behaviours, addictive behaviours ...) has been shown to be predominant in this population. However, no studies have been conducted on aspects like self-esteem, self-efficacy and extracurricular activities. In this sense, it may be interesting to match quality of life of health students in Lyon compared to the results of the other studies carried out in France, and to have a global approach of the factors influencing quality of life, with identification of factors that are potentially harmful, but also beneficial to the global health. This study will also compare the results according to the different health sectors such as medicine, pharmacy, maieutic, odontology, and sciences of rehabilitation.

Research hypothesis: the study hypothesis is that description of the quality of life and, self-efficacy, self-esteem, nutrition, anxiety, physical activity, sleep quality, and addiction parameters in health student will better characterize student's issues in order to propose an appropriate intervention to improve their global health.

The study is an observational, cross sectional and monocentric study conducted among the population of students of the Lyon 1 University in the health science field on a 9 months period.

ELIGIBILITY:
Inclusion Criteria:

* Adult (> 18 years)
* Enrolled in 3rd year of health study (Medicine, pharmacy, Institute of Rehabilitation Sciences and Techniques, odontology, maieutic) at the UCBL
* Participation at the required medical consultation at the college Health Department of UCBL

Exclusion Criteria:

* Lack of comprehension of the French language
* Implementation of protective measures
* Erasmus program

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study target the exhaustivity of the eligible population since all students are concerned by the mandatory visit.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-11 (Estimated); Primary Completion 2020-06 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Health student's quality of life: WHOQOL BREF questionnaire | Month 9
  The quality of life will be evaluated by the WHOQOL BREF questionnaire (Caria et al, 1995, Baumann et al, 2010) consisting of 26 items exploring physical health (7 items), psychological health (6 items), social relations (3 items), environment (8 items) and the quality of life related to health attesting to the overall satisfaction (2 items). Subject responses are collected using a Likert scale, scored from 1 to 5, summed and converted to a scale of 0 (poor quality of life) to 100 (good quality of life).

CONTACTS AND LOCATIONS:
Overall Officials: Julie Haesebaert, MD, Study Director — Hospices Civils de Lyon
Locations (1):
- University Health Department Lyon, Lyon, France